CLINICAL TRIAL: NCT06929377
Title: Effectiveness of a Judo-specific Injury Prevention Programme on Performance: a Randomized Controlled Trial in Judo Athletes
Brief Title: Effectiveness of a Judo-specific Injury Prevention Programme on Performance in Judo Athletes
Acronym: JUDO-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERCAN YILLI, Clinical Physical Therapist, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 03.2025fbu
Record Dates: First submitted 2025-03-27; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Injury Prevention in Sports; Sports Performance; Sports
Keywords: Judo; injury prevention; sports performance; a randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - IPPON Group (Experimental): Intervention Group will be completed the judo specific exercise programme. It's called as ''IPPON'' warm-up programme. The IPPON intervention is an injury prevention programme designed specifically to reduce injuries in judo athletes.The IPPON intervention consists of 36 exercises divided into (1), flexibility and agility, (2) balance and coordination and (3) strength and stability. Each category consisted of 12 exercises with 3 levels of difficulty. Athletes performed 4 exercises per category and thus 12 exercises at the start of the training at least two times per week.
  Interventions: Other: IPPON warm-up programme
- Control Group (No Intervention): Athletes in the control group were instructed to continue their usual warm-up and regular judo practice as warm-up prior to training or competition is standard routine in judo. The duration of the IPPON intervention was aligned with the average duration of the usual warm-up in the control groups.

INTERVENTIONS:
Other: IPPON warm-up programme — The IPPON intervention is an injury prevention programme designed specifically to reduce injuries in judo athletes. The trainer-supervised IPPON intervention mainly focuses on preventing musculoskeletal injuries of the shoulder, knee and ankle. The IPPON intervention consists of 36 exercises divided into (1) flexibility and agility, (2) balance and coordination and (3) strength and stability. Each category consisted of 12 exercises with 3 levels of difficulty. Athletes performed 4 exercises per category and thus 12 exercises at the start of the training at least two times per week.
  Arms: Intervention Group - IPPON Group

SUMMARY:
Judo is a popular international combat sport with an estimated 20 million active participants world-wide and participation in judo entails a substantial risk of injury in both elite and recreational judo. It is known that judo involves a significantly higher risk of sports per activity compared with another combat sports such as wrestling, karate, taekwondo an deven popular team sports such as football, basketball and volleyball. Therefore, preventing injuries in judo is so important and various interventions can use in this regard. These include; taping, warm-up and cool-down programs, proper technique trainings and exercise programs. Injury prevention programmes in other sports have been proven effective in reducing injury rates for elite and recreational athletes. In judo, research on exercise-based prevention is limited to the description of injury prevention programs, but the effectiveness of these programs has never been evaluated. The aim of this study is to investigate the effects of the judo-specific ''IPPON'' warm-up programs for injury prevention of judokas on performance parameters and incidence of injuries among professional judo athletes. In this study, the investigators research the Judo-Specific Special Conditioning Test and the Isometric/Dynamic Judogi Grip Strength Test will be evaluated for performance parameters. In addition, the Upper and Lower Extremity Y Balance Test will be evaluated for balance and the Upper Extremity Internal/External Rotation Strength Test and the Lower Extremity Hamstring/Quadriceps Strength Test will be evaluated for muscle strength assessment. The Turkish translation of the Oslo Trauma Research Center Overuse Questionnaire (OSTRC-O) will be used to monitor the incidence of injuries among professional judo athletes.

DETAILED DESCRIPTION:
Judo is a popular international combat sport with an estimated 20 million active participants worldwide. Judo is characterised by the combination of balance, coordination, flexibility, agility, speed and strength with the aim to incapacitate their opponent. It is demanding of the neuromuscular and physical capacity of athletes. Participation in judo entails a substantial risk of injury in both elite and recreational judo. Injury prevention programmes in other sports have been proven effective in reducing injury rates for elite and recreational athletes. In judo, research on exercise-based prevention is limited to the description of injury prevention programmes, but the effectiveness of these programmes has never been evaluated. The main objective of our study was to evaluate the effectiveness of the bottom-up developed trainer-based IPPON intervention on the performance parameters compared with the usual warm-up in judo athletes. The secondary objectives were to evaluate injury severity, injury incidence, location-specific prevalences, time loss and sudden and gradual onset injury recurrence rates. We hypothesised that the IPPON intervention would increase performance parameters and reduce the overall injury prevalences. The IPPON intervention is an injury prevention programme designed specifically to reduce injuries in judo athletes. IPPON intervention mainly focuses on preventing musculoskeletal injuries of the shoulder, knee and ankle. The IPPON intervention consists of 36 exercises divided into (1) flexibility and agility, (2) balance and coordination and (3) strength and stability. Each category consisted of 12 exercises with 3 levels of difficulty. Athletes performed 4 exercises per category and thus 12 exercises at the start of the training at least two times per week. Prior to the intervention exercises, athletes completed running exercises and falling techniques. Athletes in the control group were instructed to continue their usual warm-up and regular judo practice as warm-up prior to training or competition is standard routine in judo. The duration of the IPPON intervention was aligned with the average duration of the usual warm-up in the control groups. Although, not measured in the study procedure, the approximate duration of warm-up was 15 min in both groups. The primary outcome was the performance parameters (Judo-Specific Special Conditioning Test, Isometric/Dynamic Judogi Grip Strength Test, Upper and Lower Extremity Y Balance Test, Upper Extremity Internal/External Rotation Strength Test, Lower Extremity Hamstring/Quadriceps Strength Test) over 8 weeks of follow-up, and secondary outcome was the overall injury prevalences (injury severity, injury incidence, location-specific prevalences, time loss and sudden and gradual onset injury recurrence rates) measured with the Turkish translation of the Oslo Trauma Research Center Overuse Questionnaire (OSTRC-O) at 2 weekly intervals over 16 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age should be more than 13 years
* the asymptomatic judokas with no history of major injury or surgery in last 6 months,
* having experience in at least 3 years competitive judo,
* actively participating in competitive judo at least 1 year,
* competing at least in national level.

Exclusion Criteria:

* competing in paralympic sports,
* if they had any major injuries or surgeries in last 6 months,
* if they had any systemic, neurological or rheumatological diseases,
* being pre-pubertal stage (Tanner I) according to Tanner Scale,
* indicated their unwillingness to participate to this study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Specific Judo Fitness Test (SJFT) | 8 weeks
  The SJFT formula is based ona total of throws (TT) made in three sets (1-15 s, 2-30 s, 3-30 s) separated by a 10 s break and heart rate (HR) collected immediately after the test and after 1 min with the inversely related index as the primary outcome [6]. During each period the athlete (tori) been evaluated throws two partners (uke A and B; far from each by 6 m) as many time as possible using the ippon-seoi-nage technique. Both uke A and B should have a similar height and weight from the tori. Just after and one minute after the test heart rate is measured.
Isometric Judogi Grip Strength Test | 8 weeks
  Isometric judogi chin-up: the athletes were asked to keep their elbows flexed with their chin above the hands for as long as possible and holding time was clocked. The test was interrupted as soon as athletes were unable to maintain the initial isometric position. In this test, athletes were encouraged to maintain the position for as long as possible.
Dynamic Judogi Grip Strength Test | 8 weeks
  Dynamic judogi chin-up: the athletes were asked to stretch their elbows completely and then flex them until the chin was above the bar and repetitions of the complete exercise were counted. Only repetitions which were carried out completely were counted, and the test was interrupted as soon as athletes were no longer able to carry out the proposed exercise completely and/or gave up voluntarily. In this test, athletes were encouraged to carry out as many dynamic repetitions as possible.
Upper Extremity Y Balance Test (UQ-YBT) | 8 weeks
  UQ-YBT: All participants will be provided written instructions and then observed a demonstration performed by one of the investigators. In their socks or barefoot, the participants then assumed a pushup position with feet no greater than shoulder width apart. While maintaining the pushup position, the participant used his/her free hand to maximally reach, slowly and under control, in each of three directions Medial, Inferolateral, and Superolateral in a sequential order without the free hand touching down.
Lower Extremity Y Balance Test (LQ-YBT) | 8 weeks
  LQ-YBT: Consisted of unilateral lower extremity reaches in the ANT, PM and PL directions. After written instructions were given and the test was demonstrated by one of the instructors, the participants were asked to keep their stance heel down and hands on hips while performing each reach direction with the non-stance leg in socks or barefoot. After a one-minute rest period, the participants will be completed three formal testing trials for each of the ANT, PM, and PL directions.
Upper Extremity External/Internal Rotation (ER/IR) Muscle Strength Ratio | 8 weeks
  For the ER/IR muscle strength measurements, the Hand Held Dynamometer (Jamaar) will be placed 2 cm proximal of the processus styloideus ulnae, on the dorsal (ER strength) or ventral (IR strength) forearm during sitting position. Three repetitions of 5 seconds of maximal voluntary effort were performed using a ''make'' test (gradually increasing resistance up to maximum without ''breaking'' the subject's strength).
Lower Extremity Hamstring/Quadriceps (H/Q) Muscle Strength Ratio | 8 weeks
  Participants performed two maximal isometric repetitions intending to flex and extend the knee in each lower limb to assess isometric hamstring and quadriceps strength, respectively. Before the onset of the testing, participants performed a standardized and specific warm-up. For quadriceps, test will be performed on a custom-built bench while participants are in a seated position at 30° of knee flexion and 90° of hip flexion with stabilization straps around the thighs. For hamstring, the participant will be seated at the edge of a table with the hip and knee flexed to 90 degrees and hands gripping the sides of the table while the clinician stabilizes the dynamometer between the participant's leg and table. H/Q ratio will be calculated.

SECONDARY OUTCOMES:
Oslo Trauma Research Center Overuse Questionnaire (OSTRC-O) | 16 weeks
  The OSTRC questionnaire is about overuse injury and health problems. These questionnaires are tools for injury and illness registration with four essential questions used to assess the severity. Scores in each symptom range from 0 to 100. The range of values in each question is from 0 to 25, with 0 representing no problem and 25 representing the maximum problem level in each question. Therefore, questions 1 and 4 are scored 0-8-17-25, and questions 2 and 3 are scored 0-6-13-19-25.

CONTACTS AND LOCATIONS:
Overall Officials: SERCAN YILLI, MSc, Principal Investigator — Hacettepe University; ELIF TURGUT, Professor, Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara
  - Hacettepe University, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malliaropoulos NG, Callan M, Johnson J. Comprehensive training programme for judo players nine plus 9+: possible lower limb primary injury prevention. Muscles Ligaments Tendons J. 2014 Jul 14;4(2):262-8. eCollection 2014 Apr. No abstract available. PMID 25332945
- [Background] Kamitani T, Malliaropoulos NG, Omiya M, Otaka Y, Inoue K, Onidani N. On the way to the Tokyo Summer Olympic Games (2020). Prevention of severe head and neck injuries in judo: it's time for action. Br J Sports Med. 2017 Nov;51(22):1581-1582. doi: 10.1136/bjsports-2017-097681. Epub 2017 Aug 17. No abstract available. PMID 28818954
- [Background] von Gerhardt AL, Vriend I, Verhagen E, Tol JL, Kerkhoffs GMMJ, Reurink G. Systematic development of an injury prevention programme for judo athletes: the IPPON intervention. BMJ Open Sport Exerc Med. 2020 Sep 29;6(1):e000791. doi: 10.1136/bmjsem-2020-000791. eCollection 2020. PMID 33033621
- [Background] Pocecco E, Ruedl G, Stankovic N, Sterkowicz S, Del Vecchio FB, Gutierrez-Garcia C, Rousseau R, Wolf M, Kopp M, Miarka B, Menz V, Krusmann P, Calmet M, Malliaropoulos N, Burtscher M. Injuries in judo: a systematic literature review including suggestions for prevention. Br J Sports Med. 2013 Dec;47(18):1139-43. doi: 10.1136/bjsports-2013-092886. PMID 24255909
- [Background] von Gerhardt AL, Reurink G, Kerkhoffs GMMJ, Verhagen E, Krabben K, Mooren J, Gal JSI, Brons A, Joorse R, van den Broek B, Kemler E, Tol JL. Effectiveness of a judo-specific injury prevention programme: a randomised controlled trial in recreational judo athletes. Br J Sports Med. 2023 Apr;57(8):450-456. doi: 10.1136/bjsports-2022-105869. Epub 2023 Jan 30. PMID 36717214